CLINICAL TRIAL: NCT06171113
Title: A Phase 1, Randomised, Double Blind Placebo-controlled, First Time in Human Study to Evaluate the Safety and Pharmacokinetics of Single and Multiple Oral Doses and Food Effect of GSK4024484 in Healthy Adult Participants.
Brief Title: A Study to Investigate the Safety of GSK4024484 in Healthy Adult Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Medicines for Malaria Venture (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 218708
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Malaria, Falciparum
Keywords: First time in human; Safety; Pharmacokinetics; GSK4024484; Healthy adults; Food effect; Single oral doses; Multiple oral doses
MeSH Terms: conditions — Malaria, Falciparum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (12):
- 6 mg single ascending dose (SAD) Group (Experimental): Participants receive a 6 mg single dose of GSK4024484 or matching placebo, in a fasted state.
  Interventions: Drug: GSK4024484C; Drug: Placebo
- 12 mg SAD Group (Experimental): Participants receive a 12 mg single dose of GSK4024484 or matching placebo, in a fasted state.
  Interventions: Drug: GSK4024484C; Drug: Placebo
- 24 mg SAD Group (Experimental): Participants receive a 24 mg single dose of GSK4024484 or matching placebo, in a fasted state.
  Interventions: Drug: GSK4024484C; Drug: Placebo
- 40 mg SAD Group (Experimental): Participants receive a 40 mg single dose of GSK4024484 or matching placebo, in a fasted state.
  Interventions: Drug: GSK4024484C; Drug: Placebo
- 60 mg SAD Group (Experimental): Participants receive a 60 mg single dose of GSK4024484 or matching placebo, in a fasted state.
  Interventions: Drug: GSK4024484C; Drug: Placebo
- 80 mg SAD Group (Experimental): Participants receive a 80 mg single dose of GSK4024484 or matching placebo, in a fasted state.
  Interventions: Drug: GSK4024484C; Drug: Placebo
- Food Effect Group (Experimental): Participants receive a single study dose of either GSK4024484 or matching placebo in a fed state.
  Interventions: Drug: GSK4024484C; Drug: Placebo
- 100 mg SAD Group (Experimental): Participants receive a 100 mg single dose of GSK4024484 or matching placebo.
  Interventions: Drug: GSK4024484C; Drug: Placebo
- Optional Group (Experimental): Participants may be included in this group, to allow flexibility if the dose escalation needs modification or a dose level needs to be added or repeated.
  Interventions: Drug: GSK4024484C; Drug: Placebo
- 10 mg multiple ascending doses (MAD) Group (Experimental): Participants receive a single dose of 10 mg per day of GSK4024484 or matching placebo during 3 subsequent days (30 mg total).
  Interventions: Drug: GSK4024484C; Drug: Placebo
- 20 mg MAD Group (Experimental): Participants receive a single dose of 20 mg per day of GSK4024484 or matching placebo during 3 subsequent days (60 mg total).
  Interventions: Drug: GSK4024484C; Drug: Placebo
- 30 mg MAD Group (Experimental): Participants receive a single dose of 30 mg per day of GSK4024484 or matching placebo during 3 subsequent days (90 mg total).
  Interventions: Drug: GSK4024484C; Drug: Placebo

INTERVENTIONS:
Drug: GSK4024484C — Doses administrated orally with 240 mL of water.
Drug: Placebo — Doses administrated orally with 240 mL of water.

SUMMARY:
The primary purpose of the study is to characterise the safety of GSK4024484 in healthy participants within a controlled pharmacokinetic (PK) range.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be 18 to 60 years of age inclusive, at the time of signing the informed consent.
2. Participants who are considered healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac assessment.
3. A participant with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, or outside the normal reference range for the population being studied, may be included only if the Investigator considers, that the finding is unlikely to introduce additional risk factors for the participant and will not interfere with the study procedures or endpoints.
4. ALT (Alanine transaminase) and AST (Aspartate transaminase) within the normal range at screening.
5. Total bilirubin within the normal range unless the participant is known to have Gilbert's syndrome.
6. Body weight ≥50kg, and BMI within the range 19 to 32 kilogram per square metre (kg/m^2) inclusive.
7. Male participants and female participants who are not of child bearing potential.
8. The participant is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions.

Exclusion Criteria:

1. History or presence of cardiovascular (including hypertension), respiratory, hepatic, renal, gastrointestinal, endocrine, hematologic, or neurological disorders, capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention or interfering with the interpretation of data in the opinion of the investigator.
2. Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
3. An average weekly alcohol intake of >14 units a week within 6 months prior to the study. One unit is equivalent to 8 g of alcohol: a half-pint (~240 ml) of beer, 1 glass (125 ml) of wine or 1 (25 ml) measure of spirits.
4. QTcF (Fridericia's formula) >450 msec based on average of triplicate ECGs. The QTcF is the QT interval corrected for heart rate according to QTcF.
5. More than 100 ventricular ectopic complexes in 24 hrs by Holter screening or any other clinically significant Holter abnormalities determined by the investigator.
6. Presence or history of cardiac arrhythmias or cardiac disease or a family or personal history of long QT syndrome.
7. Heart rate <40 or >100 beats per minute (bpm).
8. Evidence of previous myocardial infarction or any clinically significant conduction abnormality such as (including but not specific to left complete bundle branch block, AV block [2nd degree or higher], WPW syndrome). Long standing RBBB is permitted.
9. Past or intended use of over-the-counter or prescription medication, including herbal medications, CBD-based products, PPIs or H2 antagonists within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is the longest) prior to dosing. Other concomitant medication may be considered on a case by case basis by the investigator in consultation with the medical monitor. Paracetamol is permitted (capped at ≤2 grams/day).
10. Participation in the study that would result in loss of blood or blood products in excess of 500 mL within a 56-day period.
11. Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day.
12. Current enrolment or past participation (within the last 30 days before planned first dose in this study) in any other clinical study involving an investigational study intervention or any other type of medical research.
13. Participants previously dosed in this study.
14. Presence of HBsAg [or HBcAb] at screening or within 3 months prior to first dose of study intervention.
15. Positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study intervention.
16. Positive hepatitis C RNA (ribonucleic acid) test result at screening or within 3 months prior to first dose of study intervention.
17. Positive pre-study drug/alcohol screen.
18. Positive HIV antibody test.
19. Carbon monoxide levels indicative of smoking or more than 10 pack year history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
20. Use of known recreational drugs or drugs of abuse.
21. Sensitivity to any of the study treatments, or components thereof, or drug or other allergy that, in the opinion of the Investigator or GSK Medical Monitor, contraindicates participation in the study.
22. A positive confirmation of COVID-19 infection according to local procedures.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2025-08-14 (Estimated); Study Completion 2025-08-14 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants reporting serious adverse events (SAEs) after single ascending doses | From the signing of the informed consent (Day -2) until the follow up contact (Day 38 +/- 3 days post dose)
  An SAE is defined as any untoward medical occurrence that results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant or an abnormal partner pregnancy outcome.
Percentage of participants reporting SAEs by severity after single ascending doses | From the signing of the informed consent (Day -2) until the follow up contact (Day 38 +/- 3 days post dose)
  Mild SAE = a type of adverse event (AE) that is usually transient and may require only minimal treatment or therapeutic intervention. The event does not generally interfere with usual activities of daily living. Moderate SAE = a type of AE that is usually alleviated with additional specific therapeutic intervention. The event interferes with usual activities of daily living, causing discomfort but poses no significant or permanent risk of harm to the research participant. Severe SAE = a type of AE that interrupts usual activities of daily living, or significantly affects clinical status, or may require intensive therapeutic intervention.
Percentage of participants reporting SAEs after multiple ascending doses | From the signing of the informed consent (Day -2) until the follow up contact (Day 40 +/- 3 days post dose)
  An SAE is defined as any untoward medical occurrence that results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant or an abnormal partner pregnancy outcome.
Percentage of participants reporting SAEs by severity after multiple ascending doses | From the signing of the informed consent (Day -2) until the follow up contact (Day 40 +/- 3 days post dose)
  Mild SAE = a type of AE that is usually transient and may require only minimal treatment or therapeutic intervention. The event does not generally interfere with usual activities of daily living. Moderate SAE = a type of AE that is usually alleviated with additional specific therapeutic intervention. The event interferes with usual activities of daily living, causing discomfort but poses no significant or permanent risk of harm to the research participant. Severe SAE = a type of AE that interrupts usual activities of daily living, or significantly affects clinical status, or may require intensive therapeutic intervention.
Percentage of participants reporting non-serious AEs after single ascending doses | From study dose administration (Day 1) until the follow up contact (Day 38 +/- 3 days post dose)
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention.
Percentage of participants reporting non-serious AEs by severity after single ascending doses | From study dose administration (Day 1) until the follow up contact (Day 38 +/- 3 days post dose)
  Mild AE = a type of AE that is usually transient and may require only minimal treatment or therapeutic intervention. The event does not generally interfere with usual activities of daily living. Moderate AE = a type of AE that is usually alleviated with additional specific therapeutic intervention. The event interferes with usual activities of daily living, causing discomfort but poses no significant or permanent risk of harm to the research participant. Severe AE = a type of AE that interrupts usual activities of daily living, or significantly affects clinical status, or may require intensive therapeutic intervention.
Percentage of participants reporting non-serious AEs after multiple ascending doses | From first study dose administration (Day 1) until the follow up contact (Day 40 +/- 3 days post dose)
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention.
Percentage of participants reporting non-serious AEs by severity after multiple ascending doses | From first study dose administration (Day 1) until the follow up contact (Day 40 +/- 3 days post dose)
  Mild AE = a type of AE that is usually transient and may require only minimal treatment or therapeutic intervention. The event does not generally interfere with usual activities of daily living. Moderate AE = a type of AE that is usually alleviated with additional specific therapeutic intervention. The event interferes with usual activities of daily living, causing discomfort but poses no significant or permanent risk of harm to the research participant. Severe AE = a type of AE that interrupts usual activities of daily living, or significantly affects clinical status, or may require intensive therapeutic intervention.

SECONDARY OUTCOMES:
Part A: Area under the plasma drug concentration versus time curve from time zero (pre-dose) to last time of quantifiable concentration [AUC(0-t)] of GSK4024484C following single ascending doses in fasting conditions | From study dose administration (Day 1) until the follow up contact (Day 29 +/- 1 day post dose)
Part A: Area under the plasma drug concentration versus time curve from zero (pre-dose) extrapolated to infinite time [AUC(0-∞)] of GSK4024484C following single ascending doses in fasting conditions | From study dose administration (Day 1) until the follow up contact (Day 29 +/- 1 day post dose)
Part A: Maximum observed plasma drug concentration (Cmax) of GSK4024484C following single ascending doses in fasting conditions | From study dose administration (Day 1) until the follow up contact (Day 29 +/- 1 day post dose)
Part A: Time to maximum observed plasma drug concentration (Tmax) of GSK4024484C following single ascending doses in fasting conditions | From study dose administration (Day 1) until the follow up contact (Day 29 +/- 1 day post dose)
Part A: Apparent terminal half-life (t1/2) of GSK4024484C following single ascending doses in fasting conditions | From study dose administration (Day 1) until the follow up contact (Day 29 +/- 1 day post dose)
Part B: AUC(0-t) of GSK4024484C following multiple ascending doses in fasting conditions | From first study dose administration (Day 1) until the follow up contact (Day 33 +/- 1 day post dose)
Part B: AUC(0-∞) of GSK4024484C following multiple ascending doses in fasting conditions | From first study dose administration (Day 1) until the follow up contact (Day 33 +/- 1 day post dose)
Part B: Cmax of GSK4024484C following multiple ascending doses in fasting conditions | From first study dose administration (Day 1) until the follow up contact (Day 33 +/- 1 day post dose)
Part B: Tmax of GSK4024484C following multiple ascending doses in fasting conditions | From first study dose administration (Day 1) until the follow up contact (Day 33 +/- 1 day post dose)
Part B: t1/2 of GSK4024484C following multiple ascending doses in fasting conditions | From first study dose administration (Day 1) until the follow up contact (Day 33 +/- 1 day post dose)
Part B: Area under the plasma drug concentration versus time curve from zero to time of trough plasma concentration [AUC(0-tau)] of GSK4024484C following multiple ascending doses in fasting conditions | Part B: From first study dose administration (Day 1) until the follow up contact (Day 33 +/- 1 day post dose)
Part B: Trough plasma concentration (Ctau) of GSK4024484C following multiple ascending doses in fasting conditions | From first study dose administration (Day 1) until the follow up contact (Day 33 +/- 1 day post dose)
Part A: AUC(0-t) of GSK4024484C following single ascending doses in fed conditions | From study dose administration (Day 1) until the follow up contact (Day 29 +/- 1 day post dose)
Part A: AUC(0-∞) of GSK4024484C following single ascending doses in fed conditions | From study dose administration (Day 1) until the follow up contact (Day 29 +/- 1 day post dose)
Part A: Cmax of GSK4024484C following single ascending doses in fed conditions | From study dose administration (Day 1) until the follow up contact (Day 29 +/- 1 day post dose)
Part A: Tmax of GSK4024484C following single ascending doses in fed conditions | From study dose administration (Day 1) until the follow up contact (Day 29 +/- 1 day post dose)
Part A: t1/2 of GSK4024484C following single ascending doses in fed conditions | From study dose administration (Day 1) until the follow up contact (Day 29 +/- 1 day post dose)
Part B: Observed accumulation ratio (R) of GSK4024484 based on AUC(Ro) following multiple ascending doses | At Day 1 and at Day 3
Part B: Observed accumulation ratio (R) of GSK4024484 based on Cmax(RCmax) following multiple ascending doses | At Day 1 and at Day 3

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Unit Cambridge (Cuc)-Cambridge-United Kingdom-C, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/